CLINICAL TRIAL: NCT02865239
Title: Feasibility Study of Breast MRI in Decubitus Position
Acronym: EFIMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de Cancérologie de Lorraine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015-A00578-41
Record Dates: First submitted 2016-07-05; First posted 2016-08-12 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Breast Cancer
Keywords: Imaging, Three-Dimensional; Magnetic Resonance Imaging/methods*; Breast Neoplasms/diagnosis*; Prone Position; Prospective Studies
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Patient Positioning; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supine position (Placebo Comparator): 3.0 tesla MRI in supine position
  Interventions: Procedure: Position for the 3.0 Tesla in Magnetic Resonance Imaging
- Prone position (Active Comparator): 3.0 tesla MRI in prone position
  Interventions: Procedure: Position for the 3.0 Tesla in Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Position for the 3.0 Tesla in Magnetic Resonance Imaging — Eligible patients will have a standard MRI in prone position. At the end of this examination, all patients will have an other standard MRI in supine position.
  This examination is then extended by 10 minutes without additional injection of contrast medium

SUMMARY:
Breast MRI is performed in prone position which causes a number of questions. Indeed, the correlation with mammography and echography and the identification of preoperative lesions can be complex as echography and surgery are carried in supine position while mammography is performed in standing position.

Moreover, the prone position is often considered as uncomfortable by the patients. However, there is few publications in the literature on breast MRI in decubitus position.

ELIGIBILITY:
Inclusion Criteria:

* Patient to benefit a MRI in the assessment for a breast carcinoma or a suspicious of breast carcinoma
* Assessment on 3.0 Tesla in Magnetic Resonance Imaging
* Age >18 years old
* ECOG performance status ≤ 3
* Ability to provide written informed consent form

Exclusion Criteria:

* Age < 18 years old
* Claustrophobia
* Contraindication to the injection of contrast medium Gadoline
* Contraindication to MRI
* Persons deprived of liberty or under supervision

Max Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

PRIMARY OUTCOMES:
Percentage of lesions where the topography is discordant between the positions (prone and supine). | 1 day
  The topography is considered discordant if the location of the lesion is different between prone and supine positions (location will be described as the positions on a clock) and / or the distance from the nipple to the lesion is greater than 2cm between prone and supine positions.

SECONDARY OUTCOMES:
Comfort patient in supine position compared to the prone position using a self-administered questionnaire | 1 day
distance from the anterior border of the lesion to the nipple in supine position compared to the prone position | 1 day
distance from cutaneous projection of the lesion to the nipple in supine position compared to the prone position | 1 day
distance from lesion to pectoralis major muscle in supine position compared to the prone position | 1 day
Quandrant of the lesions and positions on a clock in supine position compared to the prone position | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: OLDRINI GUILLAUME, MD, Principal Investigator — Institut de Cancérologie de Lorraine
Locations (1):
- Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy, France